CLINICAL TRIAL: NCT02796027
Title: BRIDGE: Improving HIV Service Delivery for People Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nabila El-Bassel, PhD, Professor, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAQ0952; 1R01DA041063-01 (NIH)
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2021-07

CONDITIONS: Human Immunodeficiency Virus; Substance Abuse, Intravenous
Keywords: Health Services Research
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance Abuse, Intravenous

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: BRIDGE (Experimental): NSPs assigned to this arm would receive an integrated HIV service model
  Interventions: Other: BRIDGE
- Pre-implementation (No Intervention): NSPs assigned to this arm would receive standard care (treatment as usual) and would not be exposed to the integrated HIV service model.

INTERVENTIONS:
Other: BRIDGE — BRIDGE, enhanced HIV service integration package, has three components:
  1. peer driven recruitment using a Social Network Strategy (SNS) -- which has been designated as a "high impact and highly effective" strategy by the CDC for reaching out and engaging PWID in HIV testing
  2. HCT using CTR with Rapid Testing
  3. ARTAS -- a CDC case management strategy for linking HIV-positive PWID to HIV care that addresses specific barriers and gaps in HIV service delivery in NSPs
  Other Names: Enhanced HIV service integration package
  Arms: Experimental: BRIDGE

SUMMARY:
Scaling up integrated, cost-efficient HIV services for people who inject drugs (PWID) in Needle Syringe Programs (NSPs) is urgently needed in Kazakhstan, where only one-third of the estimated 19,000 HIV-positive PWID are ever linked to HIV care and only 10% initiate ART with 4% achieving viral suppression. The study's aim is to evaluate the implementation, effectiveness, and sustainability of an integrated HIV service model in 24 NSPs located in 3 Kazakhstani city areas. This model will employ highly effective strategies that will include peer-driven recruitment of PWID in NSPs using social network strategies (SNS), integrating rapid HIV testing in NSPs with HIV Care Clinic nurses, and linking HIV positive PWID in NSPs to HIV care using the ARTAS (Anti-Retroviral Treatment and Access to Services) case management model. Findings will have important public health implications for improving HIV service delivery for PWID in the Central Asian region and other countries with injection driven epidemics.

DETAILED DESCRIPTION:
The study is designed to evaluate the implementation and effectiveness of an enhanced HIV service integration package (BRIDGE) that may be scaled up in Kazakhstan's vast network of needle-syringe programs (NSPs) for PWID. This package includes low threshold strategies of peer-driven recruitment, HIV counseling and rapid testing (HCT) in NSPs conducted by HIV care clinic nurses, and ARTAS, Centers for Disease Control and Prevention's highly effective case management strategies for linking PWID to HIV care. BRIDGE is systematically designed to address specific service barriers to testing PWID for HIV, linking them to HIV care, and promoting ART (antiretroviral therapy) initiation. This study will employ an innovative stepped wedge design to evaluate implementation and effectiveness of BRIDGE on increasing engagement in the HIV care continuum in 24 NSPs located in 3 geographically disparate Kazakhstani city areas using site-level data collected from NSPs and HIV clinics. Investigators will conduct a longitudinal panel study with a random sample of HIV-positive PWID (N=600) from three regions in Kazakhstan using repeated assessments at baseline, 6-, and 12-months follow-up. This study will employ mixed methods to identify multi-level structural, community, and organizational factors that influence the implementation and effectiveness of BRIDGE and the cost of BRIDGE, examining implications for cost-effectiveness, feasibility of expansion, and sustainability. The study builds on the investigative team's extensive HIV intervention research among PWID in Kazakhstan in collaboration with the Republican AIDS Center over the past decade. It addresses implementation research questions to improve and integrate HIV service delivery systems for PWID that are not only important to the region, but have relevance to other countries that have concurrent injection drug use and HIV epidemics.

ELIGIBILITY:
Inclusion Criteria:

* positive confirmatory HIV test;
* aged 18 or older;
* report injecting any drug in the past 30 days; and
* have had one or more contacts with NSP staff at one of the 24 NSPs

Exclusion Criteria:

* show evidence of significant psychiatric or cognitive impairment that would limit effective participation as confirmed during informed consent;
* are not fluent in Russian or Kazakh as determined during informed consent; or
* have been previously screened for or enrolled in the study confirmed by fingerprint scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Number of PWID who attend Needle Syringe Programs (NSPs) (Effectiveness Outcome) | 6 months
  NSP attendance from electronic case records
Number of PWID who receive an HIV test (Effectiveness Outcome) | 6 months
  HIV rapid testing
Number of HIV positive PWID who are referred to HIV care from NSPs (Effectiveness Outcome) | 6 months
  HIV care linkage from electronic case records

SECONDARY OUTCOMES:
Number of HIV positive NSP clients who register at HIV care clinic (Effectiveness Outcome) | 6-months
  Receipt of HIV care medical services confirmed by electronic health records
Number of HIV positive NSP clients who have a viral load <1500 (Effectiveness Outcome) | 6 months
  Viral load suppression confirmed by electronic health records
Number of HIV positive NSP clients who initiate ART (Effectiveness Outcome) | 6 months
  ART initiation confirmed by electronic health records

OTHER OUTCOMES:
Incremental cost per participant who receives HIV-related medical services (Cost-Effectiveness Outcome) | 6 months
  Costs measured from staff time records, clinical and participant records, and overhead from standard program records/reports, multiplied by published labor rates and service charges
Implementation outcomes | 6 months
  Fidelity

CONTACTS AND LOCATIONS:
Overall Officials: Nabila El-Bassel, PhD, Principal Investigator — Columbia University
Locations (2):
- Columbia University School of Social Work, New York, New York, United States
- Global Health Research Center of Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Bassel N, McCrimmon T, Wu E, Chang M, Terlikbayeva A, Hunt T, Darisheva M, Primbetova S, Davis A, Metsch LR, Feaster DJ, Baiserkin B, Abishev A, Denebayeva A, Sagimbayev B, Kurmetova K, Mashirov K, Gilbert L. Effectiveness of an Intervention to Improve HIV Service Delivery for People Who Inject Drugs in Kazakhstan: A Cluster Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244734. doi: 10.1001/jamanetworkopen.2022.44734. PMID 36454567
- [Derived] McCrimmon T, Gilbert L, Hunt T, Terlikbayeva A, Wu E, Darisheva M, Primbetova S, Kuskulov A, Davis A, Dasgupta A, Schackman BR, Metsch LR, Feaster DJ, Baiserkin B, El-Bassel N. Improving HIV service delivery for people who inject drugs in Kazakhstan: study protocol for the Bridge stepped-wedge trial. Implement Sci. 2019 Jun 14;14(1):62. doi: 10.1186/s13012-019-0909-z. PMID 31200757